CLINICAL TRIAL: NCT07045337
Title: Enhancing the Therapeutic Effect of Bracing for Adolescent Idiopathic Scoliosis With a Hybrid Bracing Protocol: A Randomized-Controlled Trial
Brief Title: Enhancing the Therapeutic Effect of Bracing for Adolescent Idiopathic Scoliosis With a Hybrid Bracing Protocol
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tsz-ping Lam, Clinical Professional Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRF 14119721; 14119721 (Other Grant/Funding Number: General Research Fund, Research Grants Council (RGC), Hong Kong)
Record Dates: First submitted 2025-06-17; First posted 2025-07-01 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS)
Keywords: Adolescent Idiopathic Scoliosis; Bracing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Bracing (Experimental): Hybrid Bracing Protocol (HyBP) combining the use of daytime Underarm Brace (UAB) and a nighttime Lateral Bending Brace
  Interventions: Other: Hybrid Bracing
- Conventional fulltime underarm bracing (UAB) (Active Comparator): Conventional group uses fulltime underarm bracing (UAB)
  Interventions: Other: Conventional fulltime Underarm Bracing

INTERVENTIONS:
Other: Hybrid Bracing — Hybrid Bracing includes daytime Underarm Brace(UAB) and nighttime Lateral Bending Brace(LBB)
  Arms: Hybrid Bracing
Other: Conventional fulltime Underarm Bracing — Conventional group includes fulltime Underarm Brace (UAB) only.
  Arms: Conventional fulltime underarm bracing (UAB)

SUMMARY:
This is a prospective randomized controlled trial investigating the therapeutic effect of the Hybrid Bracing Protocol (HyBP) over the Conventional Brace in enhancing In-brace Correction (IBC) for adolescent idiopathic scoliosis(AIS).

DETAILED DESCRIPTION:
Scoliosis is a complex three-dimensional spinal deformity and AIS is the commonest with a high prevalence of 2-4%. If left untreated, AIS can progress resulting in significant health problems including back degeneration and negative body images.

Bracing, such as Underarm Brace(UAB) used in our center, is indicated for skeletally immature patients with Cobb angle>20°. Another bracing system is a nighttime Lateral Bending Brace(LBB) designed in a bending position opposite to the convexity of the curve thus resulting in its overcorrection. If AIS becomes severe despite bracing, ultra-major surgery is indicated aiming at bony fusion of the deformed segment with instrumentation. It is therefore important to maximize treatment effectiveness with bracing to control curve progression and to avoid the need for surgery. In-brace Correction(IBC) is the percentage reduction in Cobb angle with bracing.

Studies have reported IBC is an important determinant of brace effectiveness. For enhancement of IBC, we put forward the Hybrid Bracing Protocol(HyBP) combining the use of daytime UAB and nighttime LBB. To be best of our knowledge, HyBP has never been reported in the literature. Our pilot study on 8 patients treated with HyBP and 8 Cobb-matched historical controls treated with fulltime UAB showed very promising results with IBC of 42.1±22.0% and 22.1±14.9% in the HyBP and control group respectively. We therefore propose a formal prospective rater-blinded randomized controlled trial on 120 skeletally immature AIS female subjects with single thoracolumbar or lumbar curve newly prescribed with bracing. They are randomly allocated to the HyBP Group or the Conventional Brace Group (CB Group). The primary objective is to determine if the HyBP Group has better treatment effect in terms of In-brace Correction (IBC) when compared with the CB group at 3-month and 18-month after bracing. This is a 3-year study proposal representing the first phase of a project, to be followed by the second phase of the project when all subjects of the entire cohort will be assessed on curve outcome at time of completion of bracing and at 2 years post-bracing. This study will carry significant clinical impacts in that, if proven useful, the HyBP can be used for enhancement of treatment outcomes with bracing, thus preventing the scoliotic spine from deterioration and to avoid the need for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Females with AIS diagnosed after detailed clinical and radiological evaluation by an experienced orthopaedic surgeon and
2. having a single lumbar or thoracolumbar curve with Cobb angle between 20° - 40° and
3. age 10 years and older when bracing is prescribed and
4. Risser 0 to 2 and
5. either pre-menarchal or less than 1 year post-menarchal and
6. with no prior treatment for scoliosis

Exclusion Criteria:

1. presenting with associated musculoskeletal, neurological or other conditions possibly responsible for the curvature
2. with previous surgical or orthotic treatment or
3. physical or mental disability that prevent patients from complying with the bracing protocol

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
In-brace Correction (IBC) | From date of randomization, assessed up to 2 years after bracing stopped at skeletal maturity
  Although bracing is considered to be useful, its effectiveness hinges on various factors one of which is the in-brace curve correction, ie In-brace Correction (IBC). IBC is defined as the percentage of Cobb angle change during an X-ray with the brace fitted on the patient.

SECONDARY OUTCOMES:
Curve progression | From date of randomization, assessed up to 2 years after bracing stopped at skeletal maturity
  To determine if the HyBP has better treatment outcomes in terms of control of curve progression when compared with the conventional fulltime UAB
Quality of life questionnaires | From date of randomization, assessed up to 2 years after bracing stopped at skeletal maturity
  To determine if the HyBP has better outcomes when compared with the conventional fulltime UAB in terms of quality of life as assessed by SRS-22r, Spinal Appearance Questionnaire and the Brace Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Adam Yiu Chung Lau, FRCSEd (Orth), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No
Patient privacy

DOCUMENTS (1):
  • Study Protocol (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT07045337/Prot_000.pdf